CLINICAL TRIAL: NCT06999668
Title: Prospective Randomized Controlled Trial of VR Cognitive Training in Reducing Postoperative Delirium in Elderly Patients With Cerebral Small Vessel Disease Undergoing Non-Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li Zhengqian, Associate Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00006761-M20250258; TY2025014 (Other Grant/Funding Number: Peking University Golden Resources TWing Clinical Research Program)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Delirium (POD); Cerebral Small Vessel Diseases
Keywords: postoperative delirium; cerebral small vascular disease; virtual reality; cognitive function
MeSH Terms: conditions — Emergence Delirium; Cerebral Small Vessel Diseases

STUDY DESIGN:
Intervention Model Description: A third-party statistician generated the allocation sequence using R 4.3.3 with a dynamic block design (mixed block sizes of 4 and 6), stratified by study site; the randomization scheme was uploaded to the REDCap system, where patient eligibility was verified before enrollment, and upon entering patient data into REDCap, the system automatically executed the stratified randomization.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative Training Group (Experimental)
  Interventions: Device: Virtual reality cognitive function training
- Preoperative Control Group (Sham Comparator)
  Interventions: Device: Virtual scene intervention

INTERVENTIONS:
Device: Virtual reality cognitive function training — Participants will receive VR-based cognitive training over 4-5 days prior to surgery, with three daily 30-minute sessions (8:00-10:00 AM, 12:00-2:00 PM, and 5:00-7:00 PM), ensuring a total preoperative training duration ≥6 hours.
  The intervention utilizes an immersive VR environment that simulates real-world scenarios and tasks. Training modules target multiple cognitive domains, including memory, executive function, calculation, and abstract reasoning, designed as engaging, game-like activities with a gradual learning curve.
  Each participant's regimen is personalized based on baseline cognitive assessments or physician prescriptions, adhering to the "6-hour rule" for standardized efficacy evaluation. The system incorporates adaptive difficulty adjustment, dynamically modifying task complexity in response to real-time performance.
  Arms: Preoperative Training Group
Device: Virtual scene intervention — The control group will receive non-interactive VR exposure using identical equipment and session duration as the training group (3×30-minute daily sessions for 4-5 days, totaling ≥6 hours), with all interactive functions disabled to eliminate potential media-related biases (e.g., 2D/3D cognitive load differences from tablet-based interventions) and ensure between-group differences stem solely from interactive training while maintaining blinding integrity through equivalent hardware deployment.
  Arms: Preoperative Control Group

SUMMARY:
This clinical study investigates whether virtual reality (VR)-based cognitive training can help prevent postoperative delirium (POD) in elderly non-cardiac patients with pre-existing cerebral small vessel disease (CSVD). With the global aging population undergoing more surgical procedures, POD has emerged as a serious complication in surgical patients that can prolong hospital stays and increase the risk of developing Alzheimer's disease. The study utilizes an innovative VR system that combines eye-tracking cognitive assessment with interactive rehabilitation games to evaluate and train patients' cognitive function before non-cardiac and non-intracranial operations. Conducted at Peking University Third Hospital and First Hospital, this research specifically targets patients undergoing general surgery, orthopedic surgery and other non-intracranial/non-cardiac procedures to determine if this technology-based intervention can effectively reduce POD incidence in this population while exploring its underlying mechanisms. The findings could lead to a practical solution for protecting cognitive health in elderly patients undergoing routine surgical procedures during recovery

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 65 years; Preoperative MRI diagnosis of cerebral small vessel disease (CSVD); Scheduled to undergo non-cardiac, non-intracranial procedures under general anesthesia; Expected surgery duration > 2 hours; ASA physical status classification: I-III; No use of cognitive-enhancing medications within 3 months prior to surgery; Willing to participate and provide written informed consent.

Exclusion Criteria:

Contraindications to cranial MRI (e.g., cardiac pacemaker, metallic implants, etc.); Patients experiencing subjective discomfort (dizziness, nausea, vomiting) during VR device adaptation; Severe visual or auditory impairment; Severe hepatic or renal dysfunction; Pre-existing neuropsychiatric disorders (schizophrenia, epilepsy, Parkinson's disease, delirium, etc.); Inability to complete preoperative neuropsychological assessments (dementia, deaf-mutism, communication disorders); History of cerebrovascular events (stroke, transient ischemic attack, etc.) within 3 months prior to surgery; Current use of sedatives/antidepressants or history of psychoactive substance abuse/alcoholism.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postoperative delirium | From the first day to the fifth day after surgery or from the first day after surgery to before discharge
  Follow up personnel use the Confusion Assessment Method(CAM) scale to evaluate the occurrence of postoperative delirium after anesthesia surgery

SECONDARY OUTCOMES:
Changes in postoperative cognitive function | At enrollment (baseline) and on postoperative day 5 or prior to discharge (whichever occurs first).
  Trained research personnel (certified by neurologists) administer the Montreal Cognitive Assessment (MoCA) to evaluate eight cognitive domains (visuospatial ability, executive function, memory, attention, calculation, language, abstract thinking, and orientation), with total scores ranging 0-30 (normal cognition defined as ≥26).
Amplitude of Low-Frequency Fluctuation（ALFF） of brain regions | At enrollment and immediately after completion of the preoperative intervention
  Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI) was used to measure changes in brain regions activation
Fractional Amplitude of Low-Frequency Fluctuation（fALFF) of brain regions | At enrollment and immediately after completion of the preoperative intervention
  Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI) was used to measure changes in brain regions activation
Regional Homogeneity（ReHo） of brain regions | At enrollment and immediately after completion of the preoperative intervention
  Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging (BOLD-fMRI) was used to assess the synchronization of neuronal activity within brain regions

CONTACTS AND LOCATIONS:
Overall Officials: Zhengqian Li, Associate Chief Physician, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Peking university first hospital, Beijing, Beijing Municipality
  - Peking university third hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chen CC, Li HC, Liang JT, Lai IR, Purnomo JDT, Yang YT, Lin BR, Huang J, Yang CY, Tien YW, Chen CN, Lin MT, Huang GH, Inouye SK. Effect of a Modified Hospital Elder Life Program on Delirium and Length of Hospital Stay in Patients Undergoing Abdominal Surgery: A Cluster Randomized Clinical Trial. JAMA Surg. 2017 Sep 1;152(9):827-834. doi: 10.1001/jamasurg.2017.1083. PMID 28538964
- [Background] de Vries NM, Staal JB, van der Wees PJ, Adang EM, Akkermans R, Olde Rikkert MG, Nijhuis-van der Sanden MW. Patient-centred physical therapy is (cost-) effective in increasing physical activity and reducing frailty in older adults with mobility problems: a randomized controlled trial with 6 months follow-up. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):422-35. doi: 10.1002/jcsm.12091. Epub 2015 Dec 4. PMID 27239405
- [Background] Kho W, von Haefen C, Paeschke N, Nasser F, Endesfelder S, Sifringer M, Gonzalez-Lopez A, Lanzke N, Spies CD. Dexmedetomidine Restores Autophagic Flux, Modulates Associated microRNAs and the Cholinergic Anti-inflammatory Pathway upon LPS-Treatment in Rats. J Neuroimmune Pharmacol. 2022 Jun;17(1-2):261-276. doi: 10.1007/s11481-021-10003-w. Epub 2021 Aug 6. PMID 34357471
- [Background] Aranake-Chrisinger A, Avidan MS. Postoperative delirium portends descent to dementia. Br J Anaesth. 2017 Aug 1;119(2):285-288. doi: 10.1093/bja/aex126. No abstract available. PMID 28854545
- [Background] Peden CJ, Miller TR, Deiner SG, Eckenhoff RG, Fleisher LA; Members of the Perioperative Brain Health Expert Panel. Improving perioperative brain health: an expert consensus review of key actions for the perioperative care team. Br J Anaesth. 2021 Feb;126(2):423-432. doi: 10.1016/j.bja.2020.10.037. Epub 2021 Jan 4. PMID 33413977
- [Background] Jin Z, Hu J, Ma D. Postoperative delirium: perioperative assessment, risk reduction, and management. Br J Anaesth. 2020 Oct;125(4):492-504. doi: 10.1016/j.bja.2020.06.063. Epub 2020 Aug 11. PMID 32798069
- [Background] Meara JG, Leather AJ, Hagander L, Alkire BC, Alonso N, Ameh EA, Bickler SW, Conteh L, Dare AJ, Davies J, Merisier ED, El-Halabi S, Farmer PE, Gawande A, Gillies R, Greenberg SL, Grimes CE, Gruen RL, Ismail EA, Kamara TB, Lavy C, Lundeg G, Mkandawire NC, Raykar NP, Riesel JN, Rodas E, Rose J, Roy N, Shrime MG, Sullivan R, Verguet S, Watters D, Weiser TG, Wilson IH, Yamey G, Yip W. Global Surgery 2030: evidence and solutions for achieving health, welfare, and economic development. Lancet. 2015 Aug 8;386(9993):569-624. doi: 10.1016/S0140-6736(15)60160-X. Epub 2015 Apr 26. No abstract available. PMID 25924834